CLINICAL TRIAL: NCT03105791
Title: The Effect of Patient Education on Opioid Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017Abb
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Rotator Cuff Injury
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal pre-operative education (No Intervention): • Control group received normal pre-operative education regarding surgery
- Opioid usage education (Active Comparator): • The study group received formal education detailing recommended post-operative opioid usage, side effects, dependence, and addiction
  Interventions: Other: Formal education regarding opioid usage

INTERVENTIONS:
Other: Formal education regarding opioid usage — Participannts watched a 2 minute video and were given educational materials
  Arms: Opioid usage education

SUMMARY:
Prospective, randomized clinical trial investigating the use of patient education on post-operative narcotic consumption

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* clinically indicated for an arthroscopic rotator cuff repair

Exclusion Criteria:

* Patients with irreparable rotator cuff tears
* allergic or sensitivity to the study medication
* history of gastrointestinal issues
* any evidence of glenohumeral arthritis
* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Opioid Usage | 3 months
  count of total narcotic pills not taken by patients